CLINICAL TRIAL: NCT03886012
Title: Efficacy of a Transcranial Vibrating System for Mitigation of Outcomes of Migraine Associated Vertigo
Brief Title: Efficacy of a Transcranial Vibrating System for Mitigation of Migraine Associated Vertigo
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 general concerns.
Sponsor: Otolith Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OLith10401
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Dizziness; Nausea; Headache; Confusion
Keywords: Migraine Associated Vertigo
MeSH Terms: conditions — Dizziness; Nausea; Headache; Confusion

STUDY DESIGN:
Intervention Model Description: Subjects will be given the transcranial vibrating system (the Otoband) to use when they have migraine associated vertigo (MAV). The Otoband will function for up to 4 periods of 30 minutes per day, at one of two possible pre-set power levels.
  The possible power levels are A) a level deemed to be effective, or B) a placebo (ineffective) power level. On a given calendar day, the power level remains constant. The sponsor will provide Otobands with a predetermined, randomly assigned power schedule based on calendar day.
  Subjects will use the Otoband during each MAV episode. They will fill out questionnaires about associated symptoms (dizziness, nausea, headache, brain confusion) 2 & 20 minutes after using turning the Otoband on, and 20 minutes after they stop using the Otoband.
  Outcomes measured will be compared between days with device at effective versus placebo power to determine if the Otoband affects dizziness, nausea, headache and brain confusion symptoms during MAV attacks.
Who Masked: Participant, Investigator
Masking Description: Neither the subject nor the investigators in the study will know the calendar's schedule for normal or placebo power levels. At both settings, the device will be felt to vibrate, making it unlikely that participants will be able to guess which setting is effective and which is ineffective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otoband efficacy on vertigo (Experimental): Participants will be given the transcranial vibrating system (Otoband) to be used during migrane associated vertigo (MAV) attacks. Participants will be able to use the Otoband up to 4 times, 30 minutes each time, per day. The Otoband will be set to the effective power level. Participants will fill out questionnaires about 4 symptoms associated to MAV: before, during (2 and 20 minutes after turning on the Otoband) and after the session (20 minutes after the Otoband was or has stopped). The conditions evaluated will be: dizziness, nausea, headache and brain confusion.
  Participants will complete questionnaires either online using secure HIPPA-compliant webforms, or using pre-printed questionnaires, as they prefer.
  Interventions: Device: Otoband
- Otoband sham efficacy on vertigo (Sham Comparator): Participants will be given the transcranial vibrating system (Otoband) to be used during migrane associated vertigo (MAV) attacks. Participants will be able to use the Otoband up to 4 times, 30 minutes each time, per day. The Otoband will be set to an ineffective power level, serving as a placebo. Participants will fill out questionnaires about 4 symptoms associated to MAV: before, during (2 and 20 minutes after turning on the Otoband) and after the session (20 minutes after the Otoband was or has stopped). The conditions evaluated will be: dizziness, nausea, headache and brain confusion.
  Participants will complete questionnaires either online using secure HIPPA-compliant webforms, or using pre-printed questionnaires, as they prefer.
  Interventions: Device: Otoband sham

INTERVENTIONS:
Device: Otoband — The Otoband will be used by participants during migraine associated vertigo (MAV). We expect the research subjects to use the device for at least 20 minutes, with the hardware limiting any one session to a duration of 30 minutes, up to 4 times per calendar day. The Otoband will be set to the effective power level during the course of a given calendar day.
  Arms: Otoband efficacy on vertigo
Device: Otoband sham — The Otoband will be used by participants during migraine associated vertigo (MAV) for a maximum of 30 minutes, up to 4 times per calendar day. The Otoband will be set to an ineffective power level (considered a sham device) during the course of a given calendar day.
  Arms: Otoband sham efficacy on vertigo

SUMMARY:
Vertigo is among the most common symptoms associated with migraine and affects 26.5% of migraine sufferers, leading to a dramatic impact in life limiting even the most simple activities. A new device, the OtoBand, a transcranial vibrating system, has been shown to mitigate and sometimes prevent vertigo and nausea in healthy subjects. The current study aims to determine if the Otoband can treat or reduce symptoms of Migraine Associated Vertigo (MAV).

DETAILED DESCRIPTION:
Vertigo is among the most common symptoms associated with migraine and affects 26.5% of migraine sufferers. Migraine Associated Vertigo (MAV) has a dramatic impact on daily life, impacting work, relationships, and even activities of daily living. At the current time, the mainstay of therapy for migraine is pharmaceutical intervention, either acute (particularly triptans, 2) or preventative. However, this therapy has a delayed effect and can lead to a host of side effects.

In this project we examine a device that has shown promise and might be beneficial for treating or improving the course of recovery from MAV. The Otoband is a transcranial vibrating system to be placed against the skull, preferably over the mastoid bone, behind the ear. To date, the device has only been systematically tested on healthy volunteers and has shown improvement of vertigo symptoms during the use of virtual reality systems and road motion sickness.

Individuals identified at Jefferson University medical center with a history of MAV attacks will be referred to the Otolaryngology Department where their diagnosis will be confirmed and offered to enroll in the study. Participants will be able to take home an Otoband to wear when they have MAV attacks. The Otoband will be set at the effective power (proved to reduce vertigo symptoms in previous studies) and low power (proved to not impact vertigo symptoms, considered as sham device). Participants will have to assay their vertigo symptoms before, during and immediately after wearing the Otoband to evaluate the efficacy of the device.

ELIGIBILITY:
Inclusion Criteria:

Subject between the ages of 18-65 with a history of frequent Migraine Associated Vertigo (MAV) attacks as characterized by the following:

* An episode with acute onset vertigo that lasted at least 15 minutes within the previous 30 days.
* At least 5 such episodes in the past 12 months.

Exclusion Criteria:

1. History of head injury within the last six months or currently suffering the effects of a head injury
2. Presence of severe aphasia
3. History of diagnosed neuropsychiatric disorders (e.g. hypochondriasis, major depression, schizophrenia)
4. Documented neurodegenerative disorders
5. Pregnancy [Female candidates will be asked if they are pregnant]
6. Prior disorders of hearing and balance including:

   1. Ménière's disease
   2. Multiple sclerosis
   3. Vestibular neuritis
   4. Vestibular schwannoma
   5. Sudden sensorineural hearing loss
7. History of Cerebrovascular disorders
8. History of ear operation other than myringotomy and tube placement in the past
9. Planned major surgery of the skull base (for instance, cochlear implant)
10. Systemic disorders to include chronic renal failure, cirrhosis of the liver, autoimmune disease, heart disease, lung disease, or severe arthritis
11. Individuals who cannot provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in vertigo symptoms | 2 minutes and 20 minutes after starting the Otoband; and 20 minutes after stopping the Otoband
  Questionnaire for vertigo symptoms from 0 (none) to 10 (agonizing)
Brain confusion | 2 minutes and 20 minutes after starting the Otoband; and 20 minutes after stopping the Otoband
  Questionnaire for brain confusion: scale from 0 (none) to 10 (maximum) for the 4 following symptoms: forgetful, difficulty thinking/finding words, difficulty focusing, cloudy.

SECONDARY OUTCOMES:
Change in nausea symptoms | 2 minutes and 20 minutes after starting the Otoband; and 20 minutes after stopping the Otoband
  Questionnaire for nausea symptoms from 0 (none) to 10 (agonizing)
Change in headache symptoms | 2 minutes and 20 minutes after starting the Otoband; and 20 minutes after stopping the Otoband
  Questionnaire for nausea symptoms from 0 (none) to 10 (worst pain possible)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Fitzgerald, MD, Principal Investigator — Jefferson University
Locations (1):
- Thomas Jefferson Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No